CLINICAL TRIAL: NCT03818607
Title: A Randomized, Double-Blind, Active-Controlled Phase 3 Study Evaluating the Efficacy and Safety of ABP 959 Compared With Eculizumab in Adult Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: A Study Evaluating the Efficacy and Safety of ABP 959 Compared With Eculizumab in Adult Participants With PNH
Acronym: DAHLIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150168
Record Dates: First submitted 2019-01-17; First posted 2019-01-28 (Actual); Results first posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Marchiafava-Micheli Syndrome; Paroxysmal Cold Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T (ABP 959) / R (eculizumab) (Other): ABP 959 for 52 weeks in Period 1 followed by eculizumab for 26 weeks in Period 2
  Interventions: Drug: ABP 959; Drug: Eculizumab
- R (eculizumab) / T (ABP 959) (Other): Eculizumab for 52 weeks in Period 1 followed by ABP 959 for 26 weeks in Period 2
  Interventions: Drug: ABP 959; Drug: Eculizumab

INTERVENTIONS:
Drug: ABP 959 — intravenous infusion
  Other Names: Treatment T
Drug: Eculizumab — intravenous infusion
  Other Names: Soliris; Treatment R

SUMMARY:
This is a randomized, double-blind, active-controlled phase 3 study of ABP 959 in participants with paroxysmal nocturnal hemoglobinuria.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Historical diagnosis of PNH.
* Administration of eculizumab for ≥ 6 months and currently receiving 900 mg of eculizumab.
* Hemoglobin ≥ 9.0 g/dL for at least 6 weeks before randomization.
* Lactate dehydrogenase < 1.5 × the upper limit of normal at screening.
* Platelet count ≥ 50 × 10^9/L.
* Absolute neutrophil count (ANC) ≥ 0.5 x 10^9/L (500/μL).
* Participants must be vaccinated against Neisseria meningitidis.
* Participants must sign an IRB/IEC-approved ICF before participation in any procedures.

Exclusion Criteria:

* Known or suspected hereditary complement deficiency.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure [New York Heart Association ≥ Class III], serious uncontrolled cardiac arrhythmia), peripheral vascular disease, cerebrovascular accident, or transient ischemic attack in the previous 6 months.
* Evidence of acute thrombosis (liver Doppler ultrasound of hepatic and portal veins).
* Known to be positive for human immunodeficiency virus.
* Woman who is pregnant or breastfeeding.
* Participant is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or participant is receiving other investigational agent(s).
* Participant has known sensitivity to any of the products to be administered during the study, including mammalian cell-derived drug products.
* History of meningococcal infection.
* Presence or suspicion of active bacterial infection, or recurrent bacterial infection.
* History of bone marrow transplantation.
* Red blood cell transfusion required within 12 weeks before randomization.
* Participant experienced ≥ 2 breakthrough events, (ie, signs and symptoms of intravascular hemolysis, that require dose and/or schedule adjustments of eculizumab) in the previous 12 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (24):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States
- Czechia (3):
  - Fakultní Nemocnice Brno, Brno, Jihormoravsky KRAJ
  - Fakultní Nemocnice Olomouc, Olomouc
  - Fakultní Nemocnice Ostrava, Ostrava-Poruba
- Finland (2):
  - Keski-Suomen keskussairaala Jyväskylä, Jyväskylä
  - Päijät-Häme Central Hospital, Lahti
- Hôpital Privé Sévigné, Cesson-Sévigné, Brittany Region, France
- Saint James's Hospital, Dublin, Ireland
- Italy (5):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-cesena
  - Azienda Ospedaliera San Gerardo di Monza, Monza, Monza Brianza
  - Azienda Ospedaliera S. Croce e Carle Cuneo, Cuneo
  - Azienda USL della Romagna, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Radboud Universitair Medisch Centrum, Nijmegen, Gelderland, Netherlands
- Oslo University Hospital - Rikshospitalet, Oslo, Norway
- Instituto Português de Oncologia do Porto Francisco Gentil, Porto, Portugal
- Univerzitetni klinični center Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario La Fe, Valencia
- Karolinska Universitetssjukhuset - Huddinge, Stockholm, Sweden
- Turkey (Türkiye) (2):
  - Ege Universitesi Hastanesi - Sağlık Uygulama ve Araştırma Merkezi, Bornova, İzmir
  - Mersin Universitesi Tip Fakultesi, Mersin
- United Kingdom (2):
  - The Leeds Teaching Hospitals NHS Trust, Leeds, England
  - King's College Hospital NHS Foundation Trust, London, England

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Kulasekararaj A, Lanza F, Arvanitakis A, Langemeijer S, Chonat S, Tombak A, Hanes V, Cao J, Miller MJ, Colbert A, Shander B, Mytych DT, Chow V, Henary H. Comparative clinical efficacy and safety of biosimilar ABP 959 and eculizumab reference product in patients with paroxysmal nocturnal hemoglobinuria. Am J Hematol. 2024 Nov;99(11):2108-2117. doi: 10.1002/ajh.27456. Epub 2024 Aug 22. PMID 39171864
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 25 research centers in 14 countries including the Czech Republic, Finland, France, Ireland, Italy, the Netherlands, Norway, Portugal, Slovenia, Spain, Sweden, Turkey, the United Kingdom, and the United States, and participated from 22 January 2019 to 12 July 2022
Pre-assignment Details: 42 adult participants with paroxysmal nocturnal hemoglobinuria (PNH) were enrolled and randomized in a 1:1 ratio to receive each investigational product (ABP 959 and eculizumab) in 1 of 2 treatment sequences. Randomization was stratified by red blood cell (RBC) transfusion received within the last 12 months before randomization. There was no washout between Periods 1 and 2.
Groups:
- ABP 959/Eculizumab: Participants received ABP 959 900 mg administered intravenously (IV) every 14 ± 2 days for 52 weeks in Period 1 followed by eculizumab 900 mg administered IV every 14 ± 2 days for 26 weeks in Period 2.
- Eculizumab/ABP 959: Participants received eculizumab 900 mg administered IV every 14 ± 2 days for 52 weeks in Period 1 followed by ABP 959 900 mg administered IV every 14 ± 2 days for 26 weeks in Period 2.
Period: Period 1 (Week 1 to Week 52)
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Started | 20 | 22
Participants Treated | 20 | 22
Completed | 20 | 21
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2 (Week 53 to Week 79)
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Started | 20 | 21
Participants Treated | 20 | 21
Completed | 19 | 20
Not Completed | 1 | 1
Not completed — Participant's personal needs | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ABP 959/Eculizumab: Participants received ABP 959 900 mg administered IV every 14 ± 2 days for 52 weeks in Period 1 followed by eculizumab 900 mg administered IV every 14 ± 2 days for 26 weeks in Period 2.
- Total: Total of all reporting groups
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959 | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (16.73) | 50.2 (16.90) | 50.2 (16.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 9 | 11 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 17 | 33
  Asian | 0 | 1 | 1
  Not allowed to collect | 4 | 4 | 8
RBC Transfusion Within 12 Months Before Randomization per Electronic Case Report Form (eCRF) [Count of Participants; unit: Participants]
  Yes | 2 | 3 | 5
  No | 18 | 19 | 37
Mean Number of Packed RBC Units Received in Last 12 Months [Mean (Standard Deviation); unit: Packed RBC Units] — Number of units of packed RBCs that were transfused in the 12 months prior to enrollment.
  Packed RBC Units | 1.5 (0.71) | 1.7 (1.15) | 1.6 (0.89)

OUTCOME MEASURES:

1. Primary Outcome: LDH Level at Week 27 (Parallel Comparison)
Description: The primary analysis for the parallel comparison was hemolysis as measured by LDH at Week 27 by initial treatment received (Period 1).
Time Frame: Week 27
Population: The full analysis set (FAS) included all randomized participants.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: U/L
Groups:
- ABP 959: Participants received ABP 959 900 mg administered IV every 14 ± 2 days for 52 weeks in Period 1.
- Eculizumab: Participants received eculizumab 900 mg administered IV every 14 ± 2 days for 52 weeks in Period 1.
Arm/Group | ABP 959 | Eculizumab
Number analyzed (Participants) | 20 | 22
U/L | 205.69 [191.23 to 221.24] | 193.53 [180.80 to 207.17]
Statistical Analysis 1: Comparison: ABP 959 vs Eculizumab; Test type: Non-Inferiority — The clinical similarity of the Week 27 LDH between treatments was assessed by comparing the 1-sided 97.5% upper confidence interval (CI) limit for the geometric mean ratio of LDH at Week 27 between ABP 959 treatment and eculizumab treatment with a non-inferiority margin of 2.873; Geometric LS mean ratio (GMR) = 1.0628, 97.5% CI 1-sided [upper limit 1.1576]

2. Primary Outcome: Time-adjusted Area Under the Effect Curve (AUEC) of LDH (Crossover Comparison Per Assigned Treatment)
Description: The primary analysis for the crossover comparison was hemolysis, as measured by the time-adjusted AUEC of LDH, according to treatment assigned during each of the 14-week assessments during Periods 1 and 2.
Time Frame: From Week 13 to Week 27, from Week 39 to Week 53, and from Week 65 to Week 79
Population: The modified FAS included all randomized participants with an LDH-time profile evaluable for the time-adjusted AUEC, according to treatment assigned during each of the 14-week assessments during Period 1 and 2.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: U*day/L/week
Groups:
- ABP 959: Participants who received ABP 959 900 mg in Period 1 (administered IV every 14 ± 2 days for 52 weeks) or ABP 959 900 mg in Period 2 (administered IV every 14 ± 2 days for 26 weeks).
- Eculizumab: Participants who received eculizumab 900 mg in Period 1 (administered IV every 14 ± 2 days for 52 weeks) or eculizumab 900 mg in Period 2 (administered IV every 14 ± 2 days for 26 weeks).
Arm/Group | ABP 959 | Eculizumab
Number analyzed (Participants) | 40 | 40
U*day/L/week | 1445.76 [1295.63 to 1613.28] | 1473.44 [1321.86 to 1642.41]
Statistical Analysis 1: Comparison: ABP 959 vs Eculizumab; Test type: Other — The clinical similarity of the AUEC between treatments was assessed by comparing 2-sided 90% CI for the GMR of the time-adjusted AUEC of LDH (Week 13 to Week 27, Week 39 to Week 53, and Week 65 to Week 79) between ABP 959 treatment and eculizumab treatment with a similarity margin of (0.77, 1.30); GMR = 0.9812, 90% CI 2-sided [0.9403 to 1.0239]

3. Secondary Outcome: Mean Total Complement (50% Total Hemolytic Complement Activity [CH50])
Description: Total complement (%) was measured in serum using an assay method and compared the total hemolytic complement activity to the lower limit of the normal human reference (LLN) of 58 U/mL for all CH50 values. The percent of LLN of CH50 at each time point was calculated as mean CH50 results/LLN x 100%.
  Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline, Week 27, Week 39, Week 53, Week 65, and Week 79
Population: Participants in the FAS with data available at each time point. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: Percent of LLN for all CH50 values
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
Percent of LLN for all CH50 values
  Baseline | 6.4 (13.48) | 2.6 (4.11)
  Week 27: number analyzed (Participants) | 19 | 21
  Week 27 | 7.5 (16.68) | 6.3 (12.25)
  Week 39: number analyzed (Participants) | 17 | 21
  Week 39 | 7.4 (23.80) | 5.1 (10.36)
  Week 53: number analyzed (Participants) | 20 | 21
  Week 53 | 12.0 (34.29) | 4.6 (6.84)
  Week 65: number analyzed (Participants) | 16 | 18
  Week 65 | 25.6 (65.27) | 7.8 (11.37)
  Week 79: number analyzed (Participants) | 18 | 20
  Week 79 | 15.8 (35.65) | 6.5 (12.67)

4. Secondary Outcome: Mean Total Hemoglobin Levels
Description: Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline, Week 27, Week 39, Week 53, Week 65, and Week 79
Population: Participants in the FAS with data available at each time point. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
g/L
  Baseline: number analyzed (Participants) | 20 | 21
  Baseline | 113.0 (15.03) | 113.8 (16.09)
  Week 27: number analyzed (Participants) | 18 | 20
  Week 27 | 110.6 (15.19) | 116.1 (16.08)
  Week 39: number analyzed (Participants) | 16 | 20
  Week 39 | 114.6 (14.12) | 115.0 (15.39)
  Week 53: number analyzed (Participants) | 19 | 21
  Week 53 | 109.8 (15.17) | 115.8 (15.20)
  Week 65: number analyzed (Participants) | 15 | 18
  Week 65 | 106.9 (17.74) | 115.7 (18.36)
  Week 79: number analyzed (Participants) | 19 | 20
  Week 79 | 113.0 (16.78) | 115.7 (16.75)

5. Secondary Outcome: Mean Serum-free Hemoglobin Levels
Description: Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline, Week 27, Week 39, Week 53, Week 65, and Week 79
Population: Participants in the FAS with data available at each time point. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
mg/dL
  Baseline | 9.30 (26.960) | 3.76 (2.758)
  Week 27: number analyzed (Participants) | 17 | 21
  Week 27 | 5.38 (14.839) | 3.10 (2.920)
  Week 39: number analyzed (Participants) | 17 | 21
  Week 39 | 3.74 (5.093) | 10.25 (27.926)
  Week 53: number analyzed (Participants) | 18 | 21
  Week 53 | 13.60 (33.793) | 3.08 (2.529)
  Week 65: number analyzed (Participants) | 16 | 18
  Week 65 | 3.22 (2.249) | 2.75 (2.077)
  Week 79: number analyzed (Participants) | 17 | 15
  Week 79 | 6.59 (10.232) | 13.89 (41.634)

6. Secondary Outcome: Mean Haptoglobin Levels
Description: Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline, Week 27, Week 39, Week 53, Week 65, and Week 79
Population: Participants in the FAS with data available at each time point. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
g/L
  Baseline | 0.200 (0.2562) | 0.286 (0.3714)
  Week 27: number analyzed (Participants) | 19 | 21
  Week 27 | 0.201 (0.2809) | 0.300 (0.4153)
  Week 39: number analyzed (Participants) | 18 | 21
  Week 39 | 0.196 (0.3085) | 0.301 (0.4266)
  Week 53: number analyzed (Participants) | 20 | 21
  Week 53 | 0.196 (0.2571) | 0.383 (0.6550)
  Week 65: number analyzed (Participants) | 16 | 18
  Week 65 | 0.201 (0.2521) | 0.466 (0.5624)
  Week 79: number analyzed (Participants) | 19 | 20
  Week 79 | 0.201 (0.2473) | 0.335 (0.4744)

7. Secondary Outcome: Mean Bilirubin Levels
Description: Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline, Week 27, Week 39, Week 53, Week 65, and Week 79
Population: Participants in the FAS with data available at each time point. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
micromol/L
  Baseline | 23.63 (12.537) | 21.12 (13.872)
  Week 27: number analyzed (Participants) | 19 | 21
  Week 27 | 28.69 (22.529) | 24.30 (19.209)
  Week 39: number analyzed (Participants) | 18 | 21
  Week 39 | 24.08 (14.258) | 24.15 (16.655)
  Week 53: number analyzed (Participants) | 20 | 21
  Week 53 | 25.76 (17.156) | 21.32 (14.036)
  Week 65: number analyzed (Participants) | 16 | 18
  Week 65 | 24.51 (16.736) | 20.02 (13.808)
  Week 79: number analyzed (Participants) | 19 | 20
  Week 79 | 23.73 (16.161) | 23.15 (17.286)

8. Secondary Outcome: Degree of Hemoglobinuria
Description: The degree of hemoglobinuria was categorized as negative, trace, small, moderate, and large based on the analysis of urine samples collected from each participant at the specified time points.
  Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline, Week 27, Week 39, Week 53, Week 65, and Week 79
Population: Participants in the FAS with evaluable urine samples available at each time point. The FAS included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
Participants
  Baseline: number analyzed (Participants) | 20 | 21
  Baseline: Negative | 17 | 21
  Baseline: Trace | 0 | 0
  Baseline: Small | 2 | 0
  Baseline: Moderate | 0 | 0
  Baseline: Large | 1 | 0
  Week 27: number analyzed (Participants) | 19 | 21
  Week 27: Negative | 17 | 20
  Week 27: Trace | 0 | 1
  Week 27: Small | 1 | 0
  Week 27: Moderate | 0 | 0
  Week 27: Large | 1 | 0
  Week 39: number analyzed (Participants) | 17 | 21
  Week 39: Negative | 16 | 20
  Week 39: Trace | 1 | 1
  Week 39: Small | 0 | 0
  Week 39: Moderate | 0 | 0
  Week 39: Large | 0 | 0
  Week 53: number analyzed (Participants) | 19 | 20
  Week 53: Negative | 16 | 19
  Week 53: Trace | 1 | 1
  Week 53: Small | 1 | 0
  Week 53: Moderate | 1 | 0
  Week 53: Large | 0 | 0
  Week 65: number analyzed (Participants) | 16 | 18
  Week 65: Negative | 15 | 17
  Week 65: Trace | 0 | 1
  Week 65: Small | 0 | 0
  Week 65: Moderate | 0 | 0
  Week 65: Large | 1 | 0
  Week 79: number analyzed (Participants) | 18 | 20
  Week 79: Negative | 16 | 19
  Week 79: Trace | 0 | 1
  Week 79: Small | 1 | 0
  Week 79: Moderate | 0 | 0
  Week 79: Large | 1 | 0

9. Secondary Outcome: Mean Percentage of Type III Erythrocytes
Description: As a measure of hemolysis the mean percentage of Type III erythrocytes was measured at the specified timepoints.
  Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline, Week 27, Week 39, Week 53, Week 65 and Week 79
Population: Participants in the FAS with data available at each time point. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: Percentage of Type III Erythrocytes
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
Percentage of Type III Erythrocytes
  Baseline: number analyzed (Participants) | 18 | 21
  Baseline | 39.9197 (25.36275) | 36.7478 (29.93810)
  Week 27: number analyzed (Participants) | 17 | 21
  Week 27 | 40.9121 (23.17684) | 40.1304 (30.01551)
  Week 39: number analyzed (Participants) | 16 | 20
  Week 39 | 41.2158 (24.81071) | 43.3663 (29.65777)
  Week 53: number analyzed (Participants) | 19 | 21
  Week 53 | 41.8196 (23.23819) | 40.4676 (31.14150)
  Week 65: number analyzed (Participants) | 15 | 17
  Week 65 | 39.1192 (22.20104) | 37.5379 (28.76642)
  Week 79: number analyzed (Participants) | 15 | 16
  Week 79 | 43.7609 (21.51712) | 42.5501 (30.20582)

10. Secondary Outcome: LDH Levels at Week 53 and Week 79
Description: The analysis of the crossover comparison of hemolysis, as measured by LDH at Week 53 and Week 79.
Time Frame: Week 53 (first week of Period 2) and Week 79 (last week of Period 2)
Population: Participants in the FAS with data available at each time point. The FAS included all randomized participants.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: U/L
Groups:
- ABP 959: Participants who received ABP 959 900 mg in Period 1 (administered IV every 14 ± 2 days for 52 weeks) or ABP 900 mg in Period 2 (administered IV every 14 ± 2 days for 26 weeks).
Arm/Group | ABP 959 | Eculizumab
Number analyzed (Participants) | 39 | 40
U/L | 209.95 [183.817 to 239.802] | 203.56 [178.387 to 232.295]
Statistical Analysis 1: Comparison: ABP 959 vs Eculizumab; Test type: Other; GMR = 1.0314, 97.5% CI 1-sided [upper limit 1.1201]

11. Secondary Outcome: Mean LDH Levels by Visit up to Week 79
Description: Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline, Week 3, Week 7, Week 13, Week 15, Week 19, Week 25, Week 27, Week 29, Week 33, Week 39, Week 41, Week 43, Week 45, Week 47, Week 49, Week 51, Week 53, Week 55, Week 59, Week 65, Week 67, Week 69, Week 71, Week 73, Week 75, Week 77, and Week 79
Population: Participants in the FAS with data available at each time point. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
U/L
  Baseline | 199.7 (61.06) | 193.9 (45.09)
  Week 3: number analyzed (Participants) | 19 | 20
  Week 3 | 210.7 (77.80) | 185.8 (42.22)
  Week 7: number analyzed (Participants) | 19 | 21
  Week 7 | 201.4 (48.41) | 194.0 (38.33)
  Week 13: number analyzed (Participants) | 18 | 21
  Week 13 | 207.7 (76.14) | 206.2 (63.82)
  Week 15: number analyzed (Participants) | 17 | 22
  Week 15 | 213.4 (105.86) | 197.0 (55.63)
  Week 19: number analyzed (Participants) | 19 | 21
  Week 19 | 188.5 (27.58) | 201.0 (59.21)
  Week 25: number analyzed (Participants) | 18 | 21
  Week 25 | 230.5 (76.07) | 190.2 (46.91)
  Week 27: number analyzed (Participants) | 18 | 20
  Week 27 | 191.7 (35.99) | 192.2 (63.83)
  Week 29: number analyzed (Participants) | 19 | 21
  Week 29 | 207.2 (50.35) | 202.1 (58.46)
  Week 33: number analyzed (Participants) | 17 | 20
  Week 33 | 194.6 (29.36) | 206.8 (59.44)
  Week 39: number analyzed (Participants) | 18 | 21
  Week 39 | 188.1 (37.55) | 196.9 (66.73)
  Week 41: number analyzed (Participants) | 19 | 21
  Week 41 | 196.1 (49.21) | 199.7 (51.00)
  Week 43: number analyzed (Participants) | 18 | 21
  Week 43 | 215.9 (62.41) | 207.1 (79.95)
  Week 45: number analyzed (Participants) | 19 | 21
  Week 45 | 202.8 (53.15) | 199.4 (66.14)
  Week 47: number analyzed (Participants) | 19 | 20
  Week 47 | 199.4 (51.72) | 197.6 (65.24)
  Week 49: number analyzed (Participants) | 19 | 21
  Week 49 | 216.2 (111.26) | 203.2 (68.65)
  Week 51: number analyzed (Participants) | 19 | 21
  Week 51 | 229.9 (125.47) | 197.7 (57.02)
  Week 53: number analyzed (Participants) | 20 | 21
  Week 53 | 224.0 (64.49) | 184.7 (46.32)
  Week 55: number analyzed (Participants) | 18 | 19
  Week 55 | 213.9 (103.58) | 188.0 (48.91)
  Week 59: number analyzed (Participants) | 19 | 18
  Week 59 | 209.4 (98.42) | 191.4 (79.01)
  Week 65: number analyzed (Participants) | 16 | 18
  Week 65 | 230.6 (135.26) | 180.9 (55.50)
  Week 67: number analyzed (Participants) | 19 | 17
  Week 67 | 196.1 (40.61) | 186.2 (50.57)
  Week 69: number analyzed (Participants) | 19 | 17
  Week 69 | 200.1 (38.12) | 186.2 (38.48)
  Week 71: number analyzed (Participants) | 18 | 18
  Week 71 | 196.8 (36.36) | 186.6 (48.02)
  Week 73: number analyzed (Participants) | 19 | 19
  Week 73 | 210.3 (43.90) | 181.9 (49.31)
  Week 75: number analyzed (Participants) | 17 | 19
  Week 75 | 207.9 (67.51) | 191.4 (65.08)
  Week 77: number analyzed (Participants) | 14 | 20
  Week 77 | 209.6 (54.35) | 181.4 (38.72)
  Week 79: number analyzed (Participants) | 19 | 19
  Week 79 | 229.2 (116.85) | 185.8 (45.11)

12. Secondary Outcome: Mean Number of Packed RBC Units Transfused Per Month
Description: Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Baseline to End of Study (up to Week 79)
Population: Participants in the FAS who had packed RBC units transfused. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: packed RBC units per month
Groups:
- ABP 959/Eculizumab: Participants received ABP 959 900 mg administered intravenously (IV) every 14 ± 2 days for 52 weeks in Period 1 followed by eculizumab 900 mg every 14 ± 2 days for 26 weeks in Period 2.
- Eculizumab/ABP 959: Participants received eculizumab 900 mg administered IV every 14 ± 2 days for 52 weeks in Period 1 followed by ABP 959 900 mg every 14 ± 2 days for 26 weeks in Period 2.
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 2 | 6
packed RBC units per month | 0.200 (0.1980) | 0.238 (0.2078)

13. Secondary Outcome: Total and Unbound Pharmacokinetics (PK) Area Under the Curve (AUC) of ABP 959 and Eculizumab From Week 13 to Week 15 (Period 1)
Description: The total and unbound PK concentration AUC values from Week 13 to Week 15 in Period 1 are presented by actual treatment received.
Time Frame: PK samples were collected predose and immediately postdose Week 13, 7 days post the Week 13 dose (Week 14), and predose at Week 15
Population: The PK parameter analysis set consisted of a subset of participants from the safety analysis set with an evaluable ABP 959 or eculizumab serum concentration time profile from Week 13 to Week 15.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*day/mL
Arm/Group | ABP 959 | Eculizumab
Number analyzed (Participants) | 18 | 19
µg*day/mL
  Total PK AUC | 3898.05 (37.5) | 4273.28 (30.6)
  Unbound PK AUC | 2761.19 (51.3) | 2903.93 (40.6)
Statistical Analysis 1: Comparison: ABP 959 vs Eculizumab; Total PK AUC GMR (ABP 959/Eculizumab); Test type: Other; GMR = 0.9122, 90% CI 2-sided [0.7586 to 1.0968]
Statistical Analysis 2: Comparison: ABP 959 vs Eculizumab; Unbound PK AUC GMR (ABP 959/Eculizumab); Test type: Other; GMR = 0.9508, 90% CI 2-sided [0.7454 to 1.2130]

14. Secondary Outcome: Total and Unbound Trough Serum Concentrations of ABP 959 and Eculizumab
Description: The total and unbound serum trough concentrations are presented by treatment sequence received for the prespecified time points. Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: PK samples were collected predose at the prespecified timepoints: baseline, Week 3, Week 7, Week 13, Week 15, Week 19, Week 27, Week 33, Week 39, Week 45, Week 51, Week 53, Week 55, Week 59, Week 65, Week 71, Week 77, and Week 79
Population: The PK concentration analysis set consisted of a subset of participants from the safety analysis set with at least one serum concentration (including results below the quantifiable limit) of ABP 959 or eculizumab, with data analyzed according to actual treatment received. Participants with data available at each time point are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
µg/mL
  Baseline: Total | 200.15 (52.8) | 202.58 (44.3)
  Baseline: Unbound | 94.62 (100.1) | 117.48 (71.5)
  Week 3: Total: number analyzed (Participants) | 20 | 21
  Week 3: Total | 205.25 (48.8) | 197.67 (42.9)
  Week 3: Unbound: number analyzed (Participants) | 20 | 21
  Week 3: Unbound | 113.99 (91.5) | 116.87 (68.9)
  Week 7: Total: number analyzed (Participants) | 20 | 20
  Week 7: Total | 213.51 (50.1) | 194.80 (42.5)
  Week 7: Unbound: number analyzed (Participants) | 20 | 20
  Week 7: Unbound | 116.57 (92.1) | 98.34 (108.9)
  Week 13: Total: number analyzed (Participants) | 20 | 21
  Week 13: Total | 215.54 (55.8) | 201.60 (45.6)
  Week 13: Unbound: number analyzed (Participants) | 20 | 21
  Week 13: Unbound | 114.40 (98.4) | 123.73 (69.1)
  Week 15: Total: number analyzed (Participants) | 18 | 21
  Week 15: Total | 192.80 (49.1) | 205.07 (36.9)
  Week 15: Unbound: number analyzed (Participants) | 18 | 21
  Week 15: Unbound | 98.68 (87.0) | 123.11 (66.1)
  Week 19: Total: number analyzed (Participants) | 19 | 21
  Week 19: Total | 216.46 (46.3) | 200.51 (49.1)
  Week 19: Unbound: number analyzed (Participants) | 19 | 21
  Week 19: Unbound | 133.39 (75.2) | 120.54 (77.3)
  Week 25: Total: number analyzed (Participants) | 18 | 21
  Week 25: Total | 217.75 (50.2) | 200.59 (51.7)
  Week 25: Unbound: number analyzed (Participants) | 18 | 21
  Week 25: Unbound | 134.37 (95.5) | 112.73 (96.4)
  Week 27: Total: number analyzed (Participants) | 19 | 21
  Week 27: Total | 198.17 (58.9) | 203.19 (45.3)
  Week 27: Unbound: number analyzed (Participants) | 19 | 21
  Week 27: Unbound | 112.02 (111.0) | 122.0 (83.8)
  Week 33: Total: number analyzed (Participants) | 17 | 21
  Week 33: Total | 211.62 (55.5) | 196.57 (49.1)
  Week 33: Unbound: number analyzed (Participants) | 17 | 21
  Week 33: Unbound | 130.12 (117.3) | 126.36 (78.4)
  Week 39: Total: number analyzed (Participants) | 17 | 21
  Week 39: Total | 183.57 (68.3) | 201.47 (48.1)
  Week 39: Unbound: number analyzed (Participants) | 17 | 21
  Week 39: Unbound | 131.50 (104.8) | 129.89 (75.1)
  Week 45: Total: number analyzed (Participants) | 18 | 21
  Week 45: Total | 204.62 (52.7) | 197.67 (47.9)
  Week 45: Unbound: number analyzed (Participants) | 18 | 21
  Week 45: Unbound | 130.30 (92.0) | 126.36 (77.3)
  Week 51: Total: number analyzed (Participants) | 18 | 21
  Week 51: Total | 207.20 (59.6) | 200.41 (45.5)
  Week 51: Unbound: number analyzed (Participants) | 18 | 21
  Week 51: Unbound | 130.32 (117.4) | 123.27 (68.3)
  Week 53: Total: number analyzed (Participants) | 20 | 21
  Week 53: Total | 193.77 (54.4) | 198.89 (46.3)
  Week 53: Unbound: number analyzed (Participants) | 20 | 21
  Week 53: Unbound | 108.40 (130.3) | 124.82 (74.6)
  Week 55: Total: number analyzed (Participants) | 19 | 20
  Week 55: Total | 210.22 (59.0) | 185.34 (48.4)
  Week 55: Unbound: number analyzed (Participants) | 19 | 20
  Week 55: Unbound | 132.20 (125.4) | 117.93 (77.2)
  Week 59: Total: number analyzed (Participants) | 19 | 20
  Week 59: Total | 184.38 (58.9) | 192.66 (46.6)
  Week 59: Unbound: number analyzed (Participants) | 19 | 20
  Week 59: Unbound | 111.48 (121.5) | 122.01 (78.5)
  Week 65: Total: number analyzed (Participants) | 16 | 18
  Week 65: Total | 190.09 (62.0) | 202.83 (51.5)
  Week 65: Unbound: number analyzed (Participants) | 16 | 18
  Week 65: Unbound | 110.57 (146.9) | 120.72 (87.7)
  Week 71: Total: number analyzed (Participants) | 17 | 16
  Week 71: Total | 160.43 (99.5) | 188.05 (58.6)
  Week 71: Unbound: number analyzed (Participants) | 17 | 16
  Week 71: Unbound | 101.66 (156.7) | 104.82 (115.0)
  Week 77: Total: number analyzed (Participants) | 15 | 17
  Week 77: Total | 211.80 (47.2) | 198.24 (54.8)
  Week 77: Unbound: number analyzed (Participants) | 15 | 17
  Week 77: Unbound | 140.07 (98.3) | 111.83 (99.8)
  Week 79: Total: number analyzed (Participants) | 18 | 20
  Week 79: Total | 178.29 (60.7) | 199.91 (50.0)
  Week 79: Unbound: number analyzed (Participants) | 18 | 20
  Week 79: Unbound | 101.98 (133.1) | 116.28 (96.5)

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as any adverse event (AE) that began or increased in severity or frequency at or after the time of first treatment up to end of study (up to Week 79). A treatment-emergent serious adverse event (SAE) was a TEAE that met at least 1 of the following criteria: was fatal, life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was another medically important serious event.
  The treatment-emergent events of interest (EOI) prespecified for this study included serious infections (meningococcus aspergillus, and other serious infections/sepsis), and infusion reactions.
Time Frame: Day 1 to End of Study (up to Week 79)
Population: The safety analysis set included all treated participants, with treatment assigned based on actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 959 | Eculizumab
Number analyzed (Participants) | 41 | 42
Participants
  All TEAEs | 33 | 39
  Any Treatment-emergent SAE | 7 | 2
  Any Treatment-emergent EOI: Infusion reaction | 15 | 15
  Any Treatment-emergent EOI: Serious infection | 3 | 0

16. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADAs)
Description: Any samples that tested positive for binding antibodies were also tested for neutralizing antibodies. Treatment boosted ADAs were defined as a positive immunoassay result at baseline and at least 1 postbaseline immunoassay result that was ≥ 4 times the magnitude of the baseline result. Baseline was defined as the last non-missing assessment taken prior to the first dose of IP.
Time Frame: Blood samples for ADA assessments were taken predose at baseline, Week 3, Week 7, Week 13, Week 19, Week 25, Week 27, Week 33, Week 39, Week 45, Week 51, Week 53, Week 55, Week 59, Week 65, Week 71, Week 77 and Week 79.
Population: The safety analysis set included all treated participants, with treatment assigned based on actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 959/Eculizumab | Eculizumab/ABP 959
Number analyzed (Participants) | 20 | 22
Participants
  Binding antibody positive anytime | 0 | 2
  Neutralizing antibody positive anytime | 0 | 0
  Binding antibody positive at/before baseline | 0 | 0
  Neutralizing antibody positive at/before baseline | 0 | 0
  Treatment boosted antibody positive | 0 | 0
  Binding antibody positive postbaseline with negative/no result at baseline | 0 | 2
  Overall: Neutralizing antibody positive postbaseline with negative/no result at baseline | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to End of Study (up to Week 79)
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Period 1: ABP 959: Participants received ABP 959 900 mg administered IV every 14 ± 2 days for 52 weeks in Period 1.
- Period 1: Eculizumab: Participants received eculizumab 900 mg administered IV every 14 ± 2 days for 52 weeks in Period 1.
- Period 2: ABP 959: Participants received ABP 959 900 mg administered IV every 14 ± 2 days for 26 weeks in Period 2.
- Period 2: Eculizumab: Participants received eculizumab 900 mg administered IV every 14 ± 2 days for 26 weeks in Period 2.
Arm/Group | Period 1: ABP 959 | Period 1: Eculizumab | Period 2: ABP 959 | Period 2: Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20 | 1/22 | 4/21 | 1/20
Other Adverse Events (participants affected / at risk) | 15/20 | 20/22 | 17/21 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: ABP 959 (N=20) | Period 1: Eculizumab (N=22) | Period 2: ABP 959 (N=21) | Period 2: Eculizumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vertigo CNS origin (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: ABP 959 (N=20) | Period 1: Eculizumab (N=22) | Period 2: ABP 959 (N=21) | Period 2: Eculizumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 3 | 1
Haemolysis (Blood and lymphatic system disorders) | 2 | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 1 | 0
Neovascular age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 2 | 3
Catheter site pruritus (General disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 2 | 1
Influenza like illness (General disorders) | 2 | 2 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 6 | 1 | 3 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 3 | 5
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 1 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2 | 4 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 5 | 2 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 2 | 0
Headache (Nervous system disorders) | 3 | 9 | 2 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Vertigo CNS origin (Nervous system disorders) | 1 | 0 | 0 | 0
Bilirubinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 1 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 5 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03818607/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03818607/SAP_002.pdf